CLINICAL TRIAL: NCT01858025
Title: A Pilot Feasibility Study of Definitive Concurrent Chemoradiation With Pencil Beam Scanning Proton Beam in Combination With 5-Fluorouracil and Mitomycin-C for Carcinoma of the Anal Canal
Brief Title: Concurrent Chemoradiation + 5-FU + Mitomycin-C in Anal Carcinoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jennifer Wo, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-075
Record Dates: First submitted 2013-05-16; First posted 2013-05-20 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Carcinoma of the Anal Canal
MeSH Terms: interventions — Fluorouracil; Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pencil Beam Scanning Radiation (Experimental): Pencil Beam Radiation daily, Monday-Friday, for 5-6 weeks Mitomycin-C via IV on Days 1 and 29 5-Fluorouracil via infusion pump over 4 days, starting Day 1 and 29 of chemotherapy
  Interventions: Radiation: Pencil Beam scanning Radiation; Drug: 5-fluorouracil; Drug: Mitomycin-C

INTERVENTIONS:
Radiation: Pencil Beam scanning Radiation
Drug: 5-fluorouracil
  Other Names: 5-FU
Drug: Mitomycin-C

SUMMARY:
This research study is a Pilot Study. Pilot studies are conducted to see if it is practical to do this type of research ona larger scale in the future. The pilot part of the study is to assess the possibility of using pencil beam proton radiation to treat your type of cancer. Proton radiation is used for many other types of malignancies, but its use for the treatment of anal cancer has been limited. The treatment is still being studied as research doctors are trying to find out more about its use in the treatment of anal cancer. Proton beam radiation therapy is an FDA approved radiation delivery system.

You are being asked to participate in this study because you have cancer in the anal canal. Conventional radiation therapy with photons in combination with 5-FU and mitomycin-C is used as standard treatment for many patients with anal cancer.

In this research study we are looking at another type of radiation called proton radiation, which is known to spare surrounding tissue and organs from radiation. Proton radiation delivers radiation to the area requiring radiation but delivers no dose beyond the region requiring treatment. There are several techniques that can be used to deliver proton radiation therapy. One of the newer techniques, called pencil beam scanning, allows for more accurate delivery of radiation to your tumor and further reduces the amount of normal tissue exposed to radiation. Most proton patients are treated with a number of beams that study doctors conform to the shape of your tumor. Pencil beam scanning delivers radiation with a single, narrow proton beam that is swept over the area of your tumor. This may reduce side effects that patients would normally experience with conventional radiation therapy or other means of delivering proton radiation therapy, and also minimizes treatment time.

In this research study, we are evaluating the effectiveness of using pencil beam proton radiation delivered to reduce side effects associated with radiation treatment.

DETAILED DESCRIPTION:
If you agree to participate in this study, you will be asked to undergo some screening tests or procedures to confirm that you are eligible. Many of these tests and procedures are likely to be part of regular cancer care and may be done even if it turns out that you do not take part in the research study. If you have had some of these tests or procedures recently, they may or may not have to be repeated. The screening will include the following: a medical history, physical examination, biopsy of your tumor, anal and groin exam, archival tumor tissue, CT or PET-CT, MRI, blood tests and a serum pregnancy test. If these tests show that you are eligible to participate in the research study, you will begin the study treatment. If you do not meet the eligibility criteria, you will not be able to participate in this research study.

Proton Radiation will be delivered daily for 5-6 weeks, depending on the dose prescribed by your physician. Treatment is delivered (Monday-Friday) for 5 days (no weekends or holidays). Each treatment will require that you lie on a table for 25-30 minutes.

You will receive radiation therapy as an outpatient at the Massachusetts General Hospital.

You will start receiving chemotherapy within 5 days of starting radiation treatment. The day you start chemotherapy will be considered Day 1.

You will receive Mitomycin-C on Days 1 and 29 of chemotherapy. Mitomycin-C will be delivered via IV infusion over a period of 10-30 minutes.

You will receive 5-fluorouracil on Day 1 and 29 of chemotherapy. You will be fitted with an ambulatory infusion pump that will administer 5-FU via IV infusion continuously over a period of 96 hours. The infusion pump will be about the size of a paperback book that can fit into a front-pack or "fanny-pack" around your waist. This pump will be connected to your body. The nurses in the infusion room will start the pump and disconnect it after 4 days.

At your 6 and 12 week follow up visits, a physical examination and the tests and procedures you receive will tell your study doctor whether your disease has gotten better, worse or stayed the same.

If your cancer has gotten better, you will continue to be monitored at your follow up visits.

If your cancer is suspected to have gotten worse, you will need to have a biopsy to confirm. If the biopsy is negative, you will need to come back for re-evaluation at 16 weeks (about 4 months) after completing radiation therapy.

If the biopsy confirms that your cancer has gotten worse, your doctor will recommend that you have surgery for the removal of your tumor.

If your cancer has stayed the same, your doctor will recommend that you have additional procedures done to develop a plan for treatment.

After you complete radiation therapy, you will be followed for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed invasive primary squamous, basaloid or cloacogenic carcinoma of the anal canal
* Life expectancy of at least 3 months

Exclusion Criteria:

* Prior abdominopelvic radiotherapy
* Prior systemic therapy for anal cancer
* Pregnant or breastfeeding
* Receiving other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to mitomycin-C or 5-fluorouracil
* Prior surgery for cancer of the anus that removed all macroscopic anal cancer
* Uncontrolled intercurrent illness
* AIDS based on current CDC definition
* Other immunocompromised status
* Individuals with a history of a different malignancy are ineligible except for the following circumstances: disease-free for at least 5 years or at low risk for recurrence or cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2021-11 (Actual)

PRIMARY OUTCOMES:
Feasibility of administration of pencil beam scanning proton beam radiation with chemotherapy for anal cancer | 2 years
  The primary objective of this study is to determine feasibility of administration of pencil beam scanning proton beam radiotherapy in combination with concurrent 5-fluorouracil (5-FU) and mitomycin-C for carcinoma of the anal canal. Proton radiotherapy will be considered feasible if grade 3+ skin toxicity seen on this protocol is less than 48% (reported grade 3+ dermatologic toxicity from RTOG 98-11)

SECONDARY OUTCOMES:
Assessment of Adverse Events | 2 years
  To assess rates of grade 3+ acute toxicities in the first 90 days following the start of combined modality treatment. To evaluate adverse events associated with the treatment regimens after 90 days from the start of combined modality treatment.
Quality of Life Outcomes | 2 years
  To assess health related quality-of-life outcomes after proton radiotherapy for anal carcinoma using objective measurements and validated quality-of-life instruments. Health quality of life questionnaire will be completed before treatment, within 2 weeks of completion of radiotherapy and quarterly for 15 months.
Clinical Complete Response | 12 weeks
  Estimate the clinical complete response rate at 6 weeks and 12 weeks after completion of treatment.
Radiotherapy treatment time | 2 years
  Evaluate elapsed time form radiotherapy treatment start to radiotherapy treatment end
Local-regional failure | 2 years
  Estimate the rate of local-regional failure; local-regional failure will be measured from study entry to date of first local or regional failure
Colostomy Failure and Colostomy-Free Survival | 2 years
  Estimate the rate of colostomy failure; colostomy failure will be measured from study entry to date of colostomy failure. Estimate the rate of colostomy-free survival; colostomy-free survival will be measured from study entry.
Disease-free Survival | 2 years
  Estimate the rate of disease-free survival; disease-free survival will be measured from study entry to date of first local, regional, distant or second primary failure or date of death.
Overall Survival | 2 years
  Estimate the rate of overall survival; overall survival will be measured from study entry to date of death.
Correlative Studies | 2 years
  Evaluate prevalence and prognostic significance of Bcl-2, Bcl-X1, HPV
To describe mood in the study population | 2 years
  To describe QOL and mood in this study population to help us better identify the side effects and challenges faced by patients.
To measure utilization of health services | 2 years
  To measure utilization of health services (emergency room, hospital and intensive care unit) in the study population.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Y. Wo, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Roberts Proton Therapy Center of the University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Wo JY, Plastaras JP, Metz JM, Jiang W, Yeap BY, Drapek LC, Adams J, Baglini C, Ryan DP, Murphy JE, Parikh AR, Allen JN, Clark JW, Blaszkowsky LS, DeLaney TF, Ben-Josef E, Hong TS. Pencil Beam Scanning Proton Beam Chemoradiation Therapy With 5-Fluorouracil and Mitomycin-C for Definitive Treatment of Carcinoma of the Anal Canal: A Multi-institutional Pilot Feasibility Study. Int J Radiat Oncol Biol Phys. 2019 Sep 1;105(1):90-95. doi: 10.1016/j.ijrobp.2019.04.040. Epub 2019 May 22. PMID 31128146